CLINICAL TRIAL: NCT03253848
Title: A Simplified Patient Care Strategy to Decrease Early Deaths in Acute Promyelocytic Leukemia (APL)
Brief Title: Simplified Patient Care Strategy in Decreasing Early Death in Patients With Acute Promyelocytic Leukemia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EA9131; NCI-2016-01123 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA9131 (Other: ECOG-ACRIN Cancer Research Group); EA9131 (Other: CTEP); UG1CA189828 (NIH); U10CA037403 (NIH)
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Acute Promyelocytic Leukemia With PML-RARA; t(15;17)
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simplified Patient Care Strategy plus APL Expert Support (Experimental): Patients receive standard of care treatment for APL. Treating physicians regularly discuss with an APL expert to identify and mange treatment.
  Interventions: Other: Simplified Patient Care Strategy; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Simplified Patient Care Strategy — Treatment per Acute Promyelocytic Leukemia (APL) Treatment Guidelines plus discussion between doctors and APL expert
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This clinical trial studies how well simplified patient care strategy works in decreasing early death in patients with acute promyelocytic leukemia. Implementing simplified acute promyelocytic leukemia guidelines along with support from acute promyelocytic leukemia experts may decrease deaths and improve survival.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate if the proposed patient care strategy, that includes use of simplified guidelines along with acute promyelocytic leukemia (APL) expert support, decreases the one-month induction mortality rate from 30% to under 15%.

SECONDARY OBJECTIVES:

I. To assess the overall survival 1 year after accrual is completed. II. To assess incidence and severity of differentiation syndrome. III. To correlate outcomes with time to initiation of all-trans retinoic acid (ATRA) from diagnosis or suspicion of diagnosis.

IV. To compare outcomes between academic and community centers separately. V. To evaluate factors associated with outcome.

OUTLINE:

Patients receive standard of care treatment for APL. Patients and doctors regularly discuss with an APL expert to identify and mange treatment.

After diagnosis, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed to have a diagnosis of APL, which is defined as:

  * Positive t(15:17) by fluorescence in situ hybridization (FISH) or conventional karyotype
  * Positive promyelocytic leukemia/retinoic acid receptor PML/RAR alpha by polymerase chain reaction (PCR)
* Patients must accept treatment and supportive care guidelines
* Referrals must be made as early as possible but no later than 5 calendar days after ATRA therapy is initiated; consent can be obtained up till day 7 or earlier
* Co-management can be started as soon as referral is made including weekends; the physician at the outlying facility should make every effort to call the APL expert at the first suspicion of APL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Anand Jillella, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (294):
- United States (282):
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Good Samaritan Medical Center, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - McKee Medical Center, Loveland, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Low Country Cancer Care Associates PC, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - AdventHealth Infusion Center Haywood, Clyde, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Main Line Health Center-Collegeville, Collegeville, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Main Line Health Center-Exton, Exton, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - MultiCare Auburn Medical Center, Auburn, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Lakeview Medical Center-Marshfield Clinic, Rice Lake, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
- Puerto Rico (12):
  - Advance Oncology Center, Aguadilla
  - Doctor's Cancer Center-Arecibo, Arecibo
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Hematologia Oncologia San Pablo, Bayamón
  - HIMA San Pablo Oncologic Hospital, Caguas
  - Doctors Cancer Center, Manatí
  - Instituto Oncologia Moderna Ponce, Ponce
  - San Juan Community Oncology Group, San Juan
  - Primary Care Physician Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - San Juan City Hospital, San Juan
  - Centro de Hematologia y Oncologia del Sur, Santa Isabel

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

REFERENCES:
- [Derived] Jillella AP, Lee SJ, Altman JK, Luger SM, Tallman MS, Foran JM, Bradshaw D, Law LY, Bryan LJ, Abou Zahr A, Begna KH, Perl AE, Vadakara JJL, Qamar R, Bergan RC, Fisch MJ, Carlos RC, Wagner LI, Kota VK, Litzow MR. Academic Community Partnership in Acute Promyelocytic Leukemia and Early Mortality: The ECOG-ACRIN EA9131 Trial. JAMA Oncol. 2025 Feb 27;11(4):400-7. doi: 10.1001/jamaoncol.2024.7033. Online ahead of print. PMID 40014329

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on August 16, 2017, and closed to accrual on July 2, 2021. A total of 202 patients were enrolled.
Groups:
- Simplified Patient Care Strategy plus APL Expert Support: All evaluable patients are included in this analysis.
Period: Overall Study
Arm/Group | Simplified Patient Care Strategy plus APL Expert Support
Started | 202
Evaluable patients | 201
Evaluable patients with toxicity data | 199
Completed | 184
Not Completed | 18
Not completed — Adverse Event | 7
Not completed — Death | 5
Not completed — initiation of other treatments | 3
Not completed — Other complicating disease | 1
Not completed — Withdrawal by Subject | 1
Not completed — Declining health | 1

BASELINE CHARACTERISTICS:
Population: All evaluable patients are included...
Arm/Group | Simplified Patient Care Strategy Plus APL Expert Support
Number analyzed (Participants) | 201
Age, Continuous [Median (Full Range); unit: years] | 53 [18 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36
  Not Hispanic or Latino | 161
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 23
  White | 158
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: One-month Mortality Rate
Description: Proportion of patients died within one month from the first date of induction therapy.
Time Frame: Assessed at one month
Population: All evaluable patients are included in this analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Groups:
- Simplified Patient Care Strategy plus APL Expert Support: Treatment per Acute Promyelocytic Leukemia (APL) Treatment Guidelines plus discussion between doctors and APL expert
Arm/Group | Simplified Patient Care Strategy plus APL Expert Support
Number analyzed (Participants) | 201
Proportion of participants | 0.03 [0.01 to 0.06]

2. Secondary Outcome: Survival Rate at One Year
Description: Overall survival is defined as the time from the first date of induction therapy to death or date last known alive. Proportion of patients alive at one year was estimated using the method of Kaplan and Meier.
Time Frame: Assessed at one year
Population: All evaluable patients are included in this analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Simplified Patient Care Strategy plus APL Expert Support
Number analyzed (Participants) | 201
Proportion of participants | 0.945 [0.903 to 0.969]

3. Secondary Outcome: One-month Survival Rate by Lead Academic Sites and Community Sites
Description: Proportion of patients who are alive at one month since the first date of induction therapy by lead academic sites and community sites
Time Frame: Assessed at one month
Population: All evaluable patients are included in this analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Groups:
- Patients accrued by lead academic sites: Patients accrued by the lead academic sites
- Patients accrued by community sites: Patients accrued by the community sites
Arm/Group | Patients accrued by lead academic sites | Patients accrued by community sites
Number analyzed (Participants) | 62 | 139
Proportion of participants | 0.952 [0.857 to 0.984] | 0.978 [0.935 to 0.993]

4. Secondary Outcome: Differentiation Syndrome Rate
Description: The proportion of patients with differentiation syndrome (measured based on the CTC version 4.0) will be evaluated.
Time Frame: Assessed up to 1 year
Reporting Status: Not Posted

5. Secondary Outcome: Association Between One-month Mortality Rate and Time From Diagnosis to Initiation of All-trans Retinoic Acid (ATRA)
Description: The time from diagnosis and initiation of ATRA will be assessed and dichotomized as "short' vs. "long" using the median value. One-month mortality rate will be compared in these two groups (short vs. long) using the Fisher's exact test.
Time Frame: Assessed at one month
Reporting Status: Not Posted

6. Secondary Outcome: Association Between One-month Survival and Baseline Factors
Description: The associations between one-month survival and baseline factors will be evaluated.
Time Frame: Assessed at baseline and one month
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed while on treatment and for 30 days after the end of treatment, up to 1 year
Description: All evaluable patients were included in the all-cause mortality analysis, while only patients with toxicity data were included in the adverse event analysis.
Arm/Group | Simplified Patient Care Strategy Plus APL Expert Support
All-Cause Mortality (participants affected / at risk) | 22/201
Serious Adverse Events (participants affected / at risk) | 115/199
Other Adverse Events (participants affected / at risk) | 152/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Simplified Patient Care Strategy Plus APL Expert Support (N=199)
Anemia (Blood and lymphatic system disorders) | 44
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 13
Leukocytosis (Blood and lymphatic system disorders) | 7
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 3
Ventricular arrhythmia (Cardiac disorders) | 1
Death NOS (General disorders and administration site conditions) | 4
Fatigue (General disorders and administration site conditions) | 2
Multi-organ failure (General disorders and administration site conditions) | 1
General disorders and administration site conditions - Other, specify (General disorders and administration site conditions) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 4
Immune system disorders - Other, specify (Immune system disorders) | 1
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 5
Activated partial thromboplastin time prolonged (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 19
Aspartate aminotransferase increased (Investigations) | 13
Creatinine increased (Investigations) | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 3
INR increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 15
Lymphocyte count increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 39
Platelet count decreased (Investigations) | 31
White blood cell decreased (Investigations) | 40
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2
Hyperuricemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Edema cerebral (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 3
Mania (Psychiatric disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 14
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3
Retinoic acid syndrome (Respiratory, thoracic and mediastinal disorders) | 5
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 5
Hypertension (Vascular disorders) | 7
Hypotension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Simplified Patient Care Strategy Plus APL Expert Support (N=199)
Fatigue (General disorders and administration site conditions) | 10
Non-cardiac chest pain (General disorders and administration site conditions) | 13
Alanine aminotransferase increased (Investigations) | 89
Aspartate aminotransferase increased (Investigations) | 91
Electrocardiogram QT corrected interval prolonged (Investigations) | 59
Hypocalcemia (Metabolism and nutrition disorders) | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 10
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 12
Retinoic acid syndrome (Respiratory, thoracic and mediastinal disorders) | 42
Hypertension (Vascular disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/48/NCT03253848/Prot_SAP_000.pdf